CLINICAL TRIAL: NCT05298501
Title: AMYWEB Validation Studies: Assessing Performance on Speech Tasks Via Crowdsourced Participants
Brief Title: Assessing Performance on Speech Tasks Via Crowdsourced Participants
Acronym: AMYWEB
Status: Terminated | Type: Observational
Why Stopped: Study stopped after first round of assessments and recruitment completed. Latter rounds were no longer required.
Sponsor: Novoic Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: NOV-0300
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2022-03

CONDITIONS: Cognitive Impairment; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AMYWEB-Normative: This cohort assessed over six recruitment and test phases, will be sampled to be as closely representative of the demographic population as possible.
  Interventions: Other: No intervention/exposure
- AMYWEB-Diversity: This cohort assessed over two recruitment and test phases will oversample participants from minority and mixed ethnic and racial backgrounds as well as participants from lower educational backgrounds.
  Interventions: Other: No intervention/exposure
- AMYWEB-MCI: This cohort assessed and recruited over one test phase, will include participants with a reported diagnosis of mild cognitive impairment or dementia.
  Interventions: Other: No intervention/exposure

INTERVENTIONS:
Other: No intervention/exposure — No interventions/exposures will be administered or evaluated

SUMMARY:
The purpose of the study is to examine the properties of the Automatic Story Recall Test (ASRT) and its parallel variants, as well as letter fluency and category fluency cognitive tests. Tests will be completed in crowdsourced populations, to derive normative data, and examine test properties in demographically diverse and cognitively impaired participants recruited and tested online.

DETAILED DESCRIPTION:
The AMYWEB study will validate speech tasks developed by NOVOIC in different population samples, including normative samples, samples recruited for enhanced demographic diversity, and participants with reported cognitive impairment.

Participants will be research volunteers recruited online and via crowdsourcing platforms. Six rounds of recruitment will be completed, evaluating different parallel variants of the Automatic Story Recall Task (ASRT), and fluency tasks. During each recruitment round participants will complete a speech test battery and questionnaires during one assessment (Baseline). Speech tasks will be recorded and later analyzed on Novoic's technology platform. All assessments will be fully online and remote.

ELIGIBILITY:
Inclusion Criteria:

* First language must be English
* Residing in the USA
* Willing to participate in a study investigating speech and dementia
* Able to provide informed consent
* Access to personal computing device that is capable of audio and video recording, and able to connect to the internet

Since key research questions are focused primarily on older-age speech and cognition, initial recruitment will be focused on older adult age brackets, which may be extended to younger adulthood if the desired sample sizes are not attained.

Exclusion Criteria:

* No formal exclusion criteria will apply at the point of recruitment and testing. however, participants with a reported history of neurological conditions or head injury, and current depression will be excluded from normative data development.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited online, primarily through crowdsourcing websites.
Sampling Method: Non-Probability Sample
Enrollment: 1034 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Age, sex, and education adjusted normative scores for the Automatic Story Recall Task (ASRT) test variants derived via linear regression analysis. | Baseline
  Participants will complete a story recall task (ASRT), which will be administered in triplets (3x stories) with immediate and delayed recall assessed.
  Six different test phases, recruiting different participant samples, will be completed in which six parallel ASRT triplets will be separately evaluated.
  Normative data will be generated for each test triplet.

SECONDARY OUTCOMES:
Normative data will be derived for shorter variants of the ASRT test battery derived via linear regression analysis. | Baseline
  Age, sex, and education adjusted normative scores for shorter test batteries established in the same way as the primary outcome for each distinct ASRT story triplet, using data from: 1 immediate recall, 2 immediate recalls, 3 immediate recalls, 3 immediate + 1 delayed recall, 3 immediate + 2 delayed recalls.
Age, sex, and education adjusted normative scores for the category fluency task performance derived via linear regression analysis. | Baseline
  During two of the study phases, participants will complete category fluency tests (participants will be asked to name as many Animals or Vegetables as they can within one minute).
Age, sex, and education adjusted normative scores for the letter fluency task performance derived via linear regression analysis. | Baseline
  During two of the study phases, participants will complete letter fluency tests (participants will be asked to say as many words as they can think of beginning with the letters F or S).
The effect of demographic differences on task performance will be evaluated via linear regression analysis. | Baseline
  The effects of age, sex, education and ethnicity on cognitive outcome measures will be evaluated for all cognitive tasks separately.
Demographic and cultural biases will be examined via group or pairwise comparison of transcription error rate and scoring errors on a simple reading task. | Baseline
  In data from a simple reading task evaluated in phases 1 and 2 of the study, transcription errors and automated scoring metrics will be evaluated alongside key demographic variables to test for cultural and demographic biases in automated transcription and scoring.
Performance differences in parallel ASRT variant tasks will be examined via task-wise comparison. | Baseline
  The distribution of test scores across parallel ASRT variants will be evaluated.
Area under the curve (AUC) of the receiver operating characteristic (ROC) curve of the binary classifier distinguishing between the MCI sample and the normative sample using as input the speech elicited during cognitive tasks. | Baseline
  Case control comparison of task performance between participants with AMYWEB-MCI and the AMYWEB-Normative population
Area under the curve (AUC) of the receiver operating characteristic (ROC) curve of the binary classifier distinguishing between depressed and non-depressed participants using as input the speech elicited during cognitive tasks. | Baseline
  All participants will complete the Participant Health Questionnaire (PHQ-8) self-report measure, alongside cognitive assessment. Participants will be separated into low depressive symptomatology (PHQ-8 scores<10), and high depressive symptomatology (PHQ-8 score>=10) groups.
The agreement between the PHQ-8 and the corresponding regression model predicting depressive symptomatology from speech data elicited during tasks will be evaluated. | Baseline
  All participants will complete the Participant Health Questionnaire (PHQ-8) self-report measure, alongside cognitive assessment.
  A continuous predictor of PHQ-8 score from speech data will be derived and covariation with continuous PHQ-8 scores will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Novoic Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided